CLINICAL TRIAL: NCT05804162
Title: A Thorough QTc Study Evaluating the Effect of Cagrilintide on Cardiac Repolarisation in Healthy Participants
Brief Title: A Research Study Looking at How Cagrilintide Works on the Heart Rhythm in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4672; U1111-1249-3834 (Other: World Health Organization (WHO)); 2022-002357-25 (EudraCT Number)
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — cagrilintide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cagrilintide (Arm 1) (Experimental): Participants will receive 0.6 milligrams (mg) of cagrilintide subcutaneously once weekly and the dose will be then escalated once in 2 weeks for 8 weeks until the target maintenance dose of 4.5 mg is reached followed by a 38-day post-treatment period. In addition, a single dose of moxifloxacin placebo prior to initiation of treatment and a single dose moxifloxacin placebo at the end of the treatment period will be administered orally.
  Interventions: Drug: Cagrilintide; Drug: Moxifloxacin Placebo
- Cagrilintide Placebo (Arm 2A) (Active Comparator): Participants will receive cagrilintide placebo subcutaenously once weekly. In addition, a single dose of moxifloxacin active prior to initiation of treatment and a single dose of moxifloxacin placebo at the end of the treatment period will be administered orally.
  Interventions: Drug: Cagrilintide Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Placebo
- Cagrilintide Placebo (Arm 2B) (Active Comparator): Participants will receive cagrilintide placebo subcutaneously once weekly. In addition, a single dose of moxifloxacin placebo prior to initiation of treatment and a single dose of moxifloxacin active at the end of the treatment period will be administered orally.
  Interventions: Drug: Cagrilintide Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Placebo

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive 0.6 mg subcutaneous injections of cagrilintide once weekly and the dose will be then escalated once in 2 weeks for 8 weeks until the target maintenance dose of 4.5 mg is reached followed by a 38-day post-treatment period.
  Other Names: Cagrilintide A; NNC0174-0833 A
  Arms: Cagrilintide (Arm 1)
Drug: Cagrilintide Placebo — Participants will receive cagrilintide placebo subcutaneously once weekly.
  Other Names: Cagrilintide A; NNC0174-0833 A
  Arms: Cagrilintide Placebo (Arm 2A); Cagrilintide Placebo (Arm 2B)
Drug: Moxifloxacin — Partcipants will receive a single dose of moxifloxacin orally.
  Other Names: Moxifloxacinratiopharm
  Arms: Cagrilintide Placebo (Arm 2A); Cagrilintide Placebo (Arm 2B)
Drug: Moxifloxacin Placebo — Partcipants will receive a single dose of moxifloxacin orally.

SUMMARY:
The study tests if treatment with cagrilintide delays the transmission of electrical signals in the heart compared to treatment with placebo. To confirm the sensitivity of the methodology, the drug moxifloxacin is also compared to a placebo in 2 treatment arms. Cagrilintide is being developed for the treatment of obesity and weight management. Moxifloxacin is an approved antibiotic for the treatment of bacterial illnesses. The study lasts for up to 17 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 23.0 and 29.9 kilogram per meter^2 (kg/m^2) (both inclusive) at screening.

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products, or to electrocardiogram (ECG) electrodes.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive method.
* History of seizures, epilepsy, repeated syncopes, cardiac arrest, cardiac arrhythmia or Torsades de Pointes (TdP), 2nd or 3rd degree atrioventricular (A-V) block or structural heart disease.
* Family history of long QT syndrome (either objectively diagnosed or suggested by sudden death due to cardiac causes before the age of 50 of a 1st degree relative).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Fridericia Heart Rate Corrected QT Interval (QTcF) At 12, 24, 48 and 72 Hours Post-Second Dose of Cagrilintide/Cagrilintide Placebo at the 4.5 mg Dose Level | From pre-last dose on Day 52 to 12, 24, 48 and 72 hours post-last dose on Day 55
  Measured in millisecond

SECONDARY OUTCOMES:
Change From Baseline in Fridericia Heart Rate Corrected QT Interval (QTcF) at 2, 3 and 4 Hours Post-Dose of Moxifloxacin/Moxifloxacin Placebo | Pre-dose to 2, 3 and 4 hours post-dose on Day 2 and Day 55
  Measured in millisecond
Change from Baseline in QT Interval Corrected Individually for HR (QTcI) at 12, 24, 48 and 72 Hours Post-Second Dose of Cagrilintide/Cagrilintide Placebo at the 4.5 mg Dose Level | From pre-last dose on Day 52 to 12, 24, 48 and 72 hours post-last dose on Day 55
  Measured in millisecond
Occurrence of Absolute QTcF Interval Prolongation: QTcF Interval > 450 millisecond (ms), QTcF Interval > 480 ms and QTcF Interval > 500 msB on ECG Recordings 0-72 Hours after Cagrilintide/Cagrilintide Placebo at the 4.5 mg Dose Levels | From pre-last dose on Day 52 to 72 hours post-last dose on Day 55
  Measured as count of participants
Occurrence of QTcF Interval Increases from Baseline > 30 ms and QTcF Interval Increases from Baseline > 60 ms Based on ECG Recordings 0-72 Hours after Cagrilintide/Cagrilintide Placebo at the 4.5 mg Dose Levels | From pre-last dose on Day 52 to 72 hours post-last dose on Day 55
  Measured as count of participants
Change from Baseline in QT Interval Corrected Individually for HR (QTcI) at 2, 3 and 4 Hours Post-Dose of Moxifloxacin/Moxifloxacin Placebo | Pre-dose to 2, 3 and 4 hours post-dose on Day 2 and Day 55
  Measured in millisecond

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency Dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Parexel International GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Gabe MBN, Fuhr R, Sinn A, Eliasen A, Berthelsen KK, Kuhlman AB, Baekdal TA, Nejad AB. Cagrilintide is not associated with clinically relevant QTc prolongation: A thorough QT study in healthy participants. Diabetes Obes Metab. 2024 Dec;26(12):5805-5811. doi: 10.1111/dom.15951. Epub 2024 Sep 16. PMID 39279639